CLINICAL TRIAL: NCT01553396
Title: Muscle Strength and Functional Autonomy of Normo-IGF-1 Elderly Women With Skeletal Muscle Dysfunctions
Brief Title: Muscle Strength and Functional Autonomy of Elderly Women
Status: Completed | Type: Observational
Sponsor: Euro-American Network of Human Kinetics (Other)
Responsible Party: Sponsor
Other Study IDs: 0165/2008
Record Dates: First submitted 2012-03-07; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Muscle, Ligament and Fascia Disorders

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This study shows an evaluation of the correlation between the muscle strength levels and functional autonomy of elderly women.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the correlation between the muscle strength levels and functional autonomy of elderly women with impaired muscle-skeletal system depending on the normal IGF-1 level. The target-population was composed by elderly women aged between 60 and 75 years (age: 67.79 ± 5.11 years, BMI: 28.01 ± 5.4), residents of an asylum, with IGF-1 levels within the normal values for the age (normo-IGF-1). Evaluations of the muscle strength (1-RM test) and the functional autonomy (GDLAM Protocol) in the performance of activities of daily living (ADL), and a measurement of basal serum levels of IGF-1 (Chemiluminescence method) were performed.

ELIGIBILITY:
Inclusion Criteria:

* present a muscle-skeletal dysfunction, such as osteoporosis, arthritis, tendinitis, but being able to perform their ADL without help from others;
* did not practice physical activity for at least 12 months;
* provide a normal IGF-1 level for their age;

Exclusion Criteria:

* elderly women unfit to perform the strength and functional autonomy tests for the medical assessment;

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of 123 elderly women residents of São Lucas shelter, located in Cacimba Velha, Teresina-PI, Brazil. The sample consists of 35 elderly women. The elderly participants in the study signed a written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Estélio HM Dantas, DSc, Study Chair — University Castelo Branco (Rio de Janeiro, Brazil)